CLINICAL TRIAL: NCT06014424
Title: Cannabidiol Medication Intervention Trial (CALM-IT)
Brief Title: Cannabidiol Medication Intervention Trial
Acronym: CALM-IT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Weston Brain Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 3878
Record Dates: First submitted 2023-07-24; First posted 2023-08-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study. Participants, Subsequent decision maker and investigator will be blinded to the treatment arm. Unblinding will not be allowed unless there are exceptional clinical circumstances that justify it
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD (Experimental): Participants randomized to the CBD arm will be titrated up to a maximum dose of 800 mg/day
  Interventions: Drug: CBD
- Placebo (Experimental): Participants randomized to the placebo will be titrated up to a maximum dose of 800 mg/day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CBD — Participants in this arm will receive CBD for 8 weeks during the first treatment period. They will then receive a two-week single-blind placebo washout before moving into the second 8-week treatment period, during which they will receive the opposite study treatment than the one given in the first treatment period.
  Arms: CBD
Other: Placebo — Participants in this arm will receive placebo for 8 weeks during the first treatment period. They will then receive a two-week single-blind placebo washout before moving into the second 8-week treatment period, during which they will receive the opposite study treatment than the one given in the first treatment period.
  Arms: Placebo

SUMMARY:
CALM-IT is a Randomized, double-blind, placebo-controlled cross-over clinical trial. Safety and efficacy of cannabidiol (CBD) capsules assessed for managing agitation in patients with AD and to identify novel biomarkers of agitation severity and treatment response.

DETAILED DESCRIPTION:
This study will look at whether CBD is an effective treatment for agitation in Alzheimer's disease (AD). This naturally derived CBD is highly pure (99%) and made by a manufacturer who meets Health Canada guidelines Cannabis products are legal for purchase in Canada.

Agitation is common in AD and is known to correlate with physical health problems such as falls and weight loss, AD progression, and caregiver burden. Current treatments for agitation in AD are not beneficial for everyone and there are concerns regarding their safety. Treating agitation is important in improving the quality of life of AD patients and their families and there is a need to identify safer and more effective treatments for agitation in AD.

The structure of this trial is called a "cross-over study". Participants will be randomized to receive either CBD or placebo during the first of two treatment phases. They will then cross-over to the opposite treatment during the second treatment phase. Participants will be on the study treatment for a total of 19 weeks and then will be followed for 4 more weeks after finishing the study treatment. There will be 12 study visits approximately every 2 weeks and 8 telephone visits every week during the study.

In addition to looking at the effectiveness of CBD in treating agitation, the researchers will also look at whether it is beneficial for other relevant outcomes for patients with AD including overall neuropsychiatric symptoms, caregiver distress, cognition, nutritional status, and pain.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥55 years of age; female must be post-menopausal or must agree to comply with contraception requirements. Males should also abide by contraceptive requirements when the partner is a woman of childbearing potential. Acceptable methods of contraception include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, which may be oral, intravaginal, or transdermal; progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, or implantable; intrauterine device or intrauterine hormone-releasing system; vasectomy of a female subject's male partner (with medical assessment and confirmation of vasectomy surgical success); bilateral tubal occlusion
2. Diagnostic and Statistical Manual of Mental Disorders-5 (DSM 5) criteria for Major Neurocognitive Disorder due to possible AD. Patients with Major Neurocognitive Disorder due to multiple etiologies (AD and vascular) will be included
3. sMMSE ≤24
4. Presence of clinically significant agitation based on the IPA definition at both screening and baseline
5. If treated with cognitive-enhancing medications (cholinesterase inhibitors and/or memantine), dosage must be stable for at least 3 months prior to study randomization
6. Availability of a primary caregiver to accompany the participant to study visits and to participate in the study. The primary caregiver must be sufficiently proficient in English to complete the required study assessments, as per investigator judgement and should spend at least 10 hours a week with the participant
7. Willing and able to provide informed consent and/or have a Substitute Decision Maker (SDM) provide informed consent on behalf of the participant

Exclusion Criteria:

1. Change in psychotropic medications less than the duration of 5 half-lives of the medication in question prior to screening (e.g., concomitant antidepressants or atypical antipsychotics) and any changes during study participation
2. Contraindications to CBs, e.g. allergies to cannabis and cannabis products, potential clinically important drug-drug interactions (e.g. strong CYP3A4 inducers/inhibitors, anticonvulsants)
3. Vascular disease, clinically important cerebrovascular disease or current uncontrolled cardiovascular disease (e.g. uncontrolled hypertension, ischemic heart disease, arrhythmia and severe heart failure, cardiovascular accident in the 3 months prior to Screening (V1)), as per investigator assessment
4. Clinically significant liver disease, as reflected by serum alanine aminotransferase or aspartate aminotransferase > 2 x upper limit of normal (ULN), or total bilirubin > 1.5 x ULN; The Investigator may decide to repeat the assessment to confirm criterion prior to screen failing the participant
5. Clinically significant impaired renal function at screening, as per investigator assessment
6. Currently meeting DSM 5 criteria for Major Depressive Episode Presence, or current substance dependence (excluding caffeine and nicotine) or history of other major psychiatric disorders or neurological conditions (e.g. psychotic disorders, schizophrenia, stroke, epilepsy)
7. Substance-Related Disorders (excluding caffeine and nicotine)
8. Clinically significant delusions and/or hallucinations (e.g. NPI-NH delusion/hallucinations subscore ≥4 or judgement of QI)
9. Reported use of marijuana or cannabinoid-based medications, products or supplements (botanical or synthetic) within 1 week prior to randomization
10. Systolic blood pressure (SBP) < 90 mmHg or > 150 mmHg or diastolic blood pressure (DBP) < 50mmHg or > 105 mmHg at screening or baseline (prior to randomization) or a postural drop in SBP ≥ 20 mmHg or DBP ≥ 10 mmHg at screening

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Agitation - Cohen-Mansfield Agitation Inventory (CMAI) | Baseline (0 Weeks) to 22 Weeks
  A 29-point scale that measures agitation in two dimensions, verbal and physical, each of which having two poles, aggressive and on-aggressive. Scores range from 29-203 points, with a higher score indicating a worse outcome.

SECONDARY OUTCOMES:
Behavior - Neuropsychiatric Inventory - Clinician Scale (NPI-C Agitation/NPI-NH) | Baseline (0 Weeks) to 22 Weeks
  NPI-C agitation is a widely used assessment of behaviour disturbances in dementia, including: apathy agitation, delusions, hallucinations, depression, euphoria, aberrant motor behaviour, irritability, disinhibition, anxiety, sleeping, and eating. NPI-NH is a caregiver-rated scale that is widely used to assess behavioral disturbances in dementia as well as caregiver distress. These behaviours include: delusions, hallucinations, agitation, aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep, appetite and eating disorders, and aberrant vocalizations. The frequency and severity of these symptoms are judged on a 4-point and 3-point scale, respectively. Scores range from 0-144 points, with a higher score indicating a worse outcome.
Cognition - Standardized Mini-Mental State Examination (sMMSE) | Baseline (0 Weeks) to 22 Weeks
  Measures global cognition, and assesses orientation to time and place, immediate recall, short-term verbal memory, calculation, language, and construct ability. Scores range from 0-30 points, with a lower score indicating a worse outcome.
Weight | Baseline (0 Weeks) to 22 Weeks
  Weight will be collected in kilograms. A change of 7% in weight will be considered clinically significant change.
Nutritional Status - Mini Nutritional Assessment - Short Form (MNA-SF) | Baseline (0 Weeks) to 22 Weeks
  A structured interview consisting of 6 items that categorizes patients as malnourished, at risk of malnutrition, or of normal nutritional status. Scores range from 0-14 points, with a lower score indicating a worse outcome.
Pain - Pain Assessment Checklist for Seniors with Limited Ability to Communicate - II (PACSLAC-II) | Baseline (0 Weeks) to 22 Weeks
  A 31-item observer-rated scale assessing facial expressions, activity/body movements, social/personality/mood indicators and mental status changes. Scores range form 0-31 points, with a higher score indicating a worse outcome.
Global Change - Alzheimer's Disease Cooperative Study - Clinical Global Impression of Severity/Change (ADCS-CGIS/C) | Baseline (0 Weeks) to 22 Weeks
  A commonly-used clinician-rated scale that quantifies disease severity and clinical change (worsening, no change, or improvement), based on information regarding the patient's medical history, cognition, behaviour, and function. Scores range from 1-7, with a lower score indicating a worse outcome.

OTHER OUTCOMES:
Sedation - Udvalg for Kliniske Undersøgelser (UKU) Side-Effect Rating Scale | Baseline (0 Weeks) to 22 Weeks
  Sedation will be measured using the Sleepiness/Sedation subscale of the UKU-Side Effect Rating Scale. The UKU is a clinician-rated scale that assesses the side effects psychopharmacological medications. Scores range from 0-3, with a higher score indicating more sleepiness/sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Krista L. Lanctot, PhD, Principal Investigator — Sunnybrook Research Institute; Giovanni Marotta, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Sciences, Whitby, Ontario

IPD SHARING:
Plan to Share IPD: No